CLINICAL TRIAL: NCT00668239
Title: Treatment of Diffuse Diabetic Maculopathy With Intravitreal Triamcinolone and Laser Photocoagulation: Randomized Clinical Trial With Morphological and Functional Evaluation
Brief Title: Diffuse Diabetic Maculopathy With Intravitreal Triamcinolone or Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: MIrela Jobim de Azevedo, MIrela Jobim de Azevedo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCPA-04288
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Macular Edema
Keywords: diffuse macular oedema; type 2 diabetes mellitus; laser therapy
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus, Type 2 | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Laser treatment: laser was applied to the macular region according to the modified grid technique in inverted C, preserving 500 μ of the foveolus and avascular zone, with 100μ diameter shots, energy varying from 0.2 to 0.5 joules, with a time of exposure between 0.2 and 0.4 seconds. One hundred and fifty to 200 shots were applied according to the size of the retinal area². ND YAG laser (Crystal Focus (EMERED®) was used
  Interventions: Procedure: laser therapy
- 2 (Experimental): triamcinolone as previously described
  Interventions: Drug: intravitreous triamcinolone

INTERVENTIONS:
Drug: intravitreous triamcinolone — Intravenous injection of 0.1 ml (4 mg) of triamcinolone acetate was performed through the pars plana in a surgical environment. The medication used was manipulated by the Ophthalmos chemist. This type of formulation is different from the similar American one (Kenalog ®) since it does not use a conservation agent
  Arms: 2
Procedure: laser therapy — pan fotocoaglulation by laser therapy
  Arms: 1

SUMMARY:
This study compares the use of intravitreous triamcinolone and laser therapy to treat maculopahty in patients with type 2 diabetes mellitus in a short-tem period of 6 months

DETAILED DESCRIPTION:
The purpose of this double blind randomized clinical trial was to compare the treatment of diffuse diabetic macular oedema with intravitreal triamcinolone and laser in patients with type 2 diabetes mellitus (DM), using a morphofunctional assessment. Patients with clinically significant diffuse macular oedema, previously untreated and with a macular thickness >250 μm at optical coherence tomography (OCT) were randomized for treatment with Laser or intravitreal injection of Triamcinolone acetate. Optical coherence tomography (OCT), biomicroscopy, fundoscopy, fluorescein angiography, tonometry, scotometry, visual acuity and contrast acuities were performed at 0, 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 DM, diffuse macular oedema secondary to diabetic retinopathy, seen at the Centre of Reference for Diabetic Retinopathy at Hospital de Clinicas de Porto Alegre (HCPA) and at the Ophthalmology Outpatient Clinic at HCPA,

Exclusion Criteria:

* patients with type 2 DM and previous treatment of diffuse macular oedema secondary to diabetic retinopathy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2004-09; Primary Completion 2006-04 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
diffuse macular oedema | 1, 3 and 6 months

SECONDARY OUTCOMES:
morphofunctional assessment of retina | 1,3 and 6 monts

CONTACTS AND LOCATIONS:
Overall Officials: Alberto L Gil, MD, Principal Investigator — Federal University of Health Science of Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - HOspital de Clínicas de Porto alegre, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Derived] Gil AL, Azevedo MJ, Tomasetto GG, Muniz CH, Lavinsky J. Treatment of diffuse diabetic maculopathy with intravitreal triamcinolone and laser photocoagulation: randomized clinical trial with morphological and functional evaluation. Arq Bras Oftalmol. 2011 Sep-Oct;74(5):343-7. doi: 10.1590/s0004-27492011000500007. PMID 22183994